CLINICAL TRIAL: NCT00056407
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Dutasteride 0.5 mg Administered Orally Once Daily for Four Years to Reduce the Risk of Biopsy-Detectable Prostate Cancer
Brief Title: "REDUCE" - A Clinical Research Study To Reduce The Incidence Of Prostate Cancer In Men Who Are At Increased Risk
Acronym: REDUCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARI40006
Record Dates: First submitted 2003-03-11; First posted 2003-03-13 (Estimated); Results first posted 2010-03-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Neoplasms, Prostate
Keywords: Prostate cancer prevention; prostate; BPH; enlarged prostate; PSA; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo Arm (Placebo Comparator): Eligible subjects will complete a 4-week placebo run-in followed by randomization to matched placebo in a 1:1 ratio.
  Interventions: Drug: Placebo
- dustasteride arm (Experimental): Eligible subjects will complete a 4-week placebo run-in followed by randomization to 0.5mg dutasteride in a 1:1 ratio. Randomization will be stratified by center.
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — After successful completion of the placebo run-in phase, subjects who continue to meet eligibility requirements will be randomized into the double-blind phase of the study and issued a 6-month supply of study drug. Subjects will self-administer study drug once daily dosing of 0.5mg of dutasteride orally for up to 4 years.
  Arms: dustasteride arm
Drug: Placebo — After successful completion of the placebo run-in phase, subjects who continue to meet eligibility requirements will be randomized into the double-blind phase of the study and issued a 6-month supply of study drug. Subjects will self-administer study drug once daily orally for up to 4 years.
  Arms: Placebo Arm

SUMMARY:
This 4-year study will compare how safe and effective an oral investigational medicine is (compared to placebo) in preventing the development of prostate cancer in men that are defined by the study entrance criteria as being at an increased risk for prostate cancer. Study visits to the clinic will occur every 6 months for up to 4 years (10 clinic visits), and a prostate biopsy will be performed at 2 and 4 years of treatment.

ELIGIBILITY:
Inclusion criteria:

* Informed consent to participate in study.
* Have had a single negative prostate biopsy within 6 months prior to enrollment in study.
* Have a PSA (prostate specific antigen) between 2.5 and 10 if 50-60 years of age; or a PSA between 3.0 and 10 if over age 60.
* Ability and will to participate in study for 4 years.

Exclusion criteria:

* More than one previous negative prostate biopsy.
* History of prostate cancer.
* Previous prostate surgery.
* Inability to urinate requiring the need of a catheter during the previous 2 years.
* Any condition (other than benign prostatic hypertrophy) which may result in urinary symptoms or changes in urine flow rate.
* Cancer within previous 5 years (other than basal or squamous cell cancers of the skin).
* Any unstable serious medical condition.
* Use within the past 12 months of finasteride (Proscar or Propecia), dutasteride (Avodart), testosterone, or drugs that can block the action of male hormones.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8231 (Actual)
Dates: Start 2003-03; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (744):
- United States (239):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Atherton, California
  - GSK Investigational Site, Culver City, California
  - GSK Investigational Site, Encino, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mather, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Pico Rivera, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Salinas, California
  - GSK Investigational Site, San Bernardino, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Temecula, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Westchester, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Trumbull, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Margate, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Okeechobee, Florida
  - GSK Investigational Site, Orange Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, South Daytona, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Stuart, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Roswell, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Galesburg, Illinois
  - GSK Investigational Site, Kankakee, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Gretna, Louisiana
  - GSK Investigational Site, Houma, Louisiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Ruston, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Greenbelt, Maryland
  - GSK Investigational Site, Owings Mills, Maryland
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Braintree, Massachusetts
  - GSK Investigational Site, Haverhill, Massachusetts
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Waltham, Massachusetts
  - GSK Investigational Site, Watertown, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Wocester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Reno, Nevada
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Lawrencevill, New Jersey
  - GSK Investigational Site, Marlton, New Jersey
  - GSK Investigational Site, Perth Amboy, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Elmont, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Garden City, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Orchard Park, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Charlotte, NC 28207, North Carolina
  - GSK Investigational Site, Concord, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Elyria, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Marion, Ohio
  - GSK Investigational Site, Zanesville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Poca City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Springfield, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Bryn Mawr, Pennsylvania
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Harrisburg, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Monroeville, Pennsylvania
  - GSK Investigational Site, Newton, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Rosemont, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, State College, Pennsylvania
  - GSK Investigational Site, Cranston, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, West Warwick, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Fort Pierre, South Dakota
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Texarkana, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Harrisonburg, Virginia
  - GSK Investigational Site, Mechanicsville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Graham, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Cheyenne, Wyoming
- Argentina (7):
  - GSK Investigational Site, Av Córdoba 2424, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Australia (10):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Woolloongabba, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Mentone, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Austria (2):
  - GSK Investigational Site, Innsbruck
  - GSK Investigational Site, Vienna
- GSK Investigational Site, Minsk, Belarus
- Belgium (11):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Mons
  - GSK Investigational Site, Turnhout
  - GSK Investigational Site, Wilrijk
  - GSK Investigational Site, Yvoir
- Brazil (6):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Rio de Janeiro, Rio de Janeiro
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Ribeirão Preto, São Paulo
  - GSK Investigational Site, São Paulo, São Paulo
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (31):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Fredericton, New Brunswick
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, Markham, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Niagara Falls, Ontario
  - GSK Investigational Site, North Bay, Ontario
  - GSK Investigational Site, North York, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Orillia, Ontario
  - GSK Investigational Site, Richmond Hill, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Granby, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Zagreb, Croatia
- Denmark (3):
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Middelfart
  - GSK Investigational Site, Nakskov
- GSK Investigational Site, Tallinn, Estonia
- Finland (9):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Rovaniemi
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (50):
  - GSK Investigational Site, Amiens
  - GSK Investigational Site, Arcachon
  - GSK Investigational Site, Auch
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bois-Bernard
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Boujan-sur-Libron
  - GSK Investigational Site, Cabestany
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Carpentras
  - GSK Investigational Site, Chalon-sur-Saône
  - GSK Investigational Site, Châlons-en-Champagne
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Domarin
  - GSK Investigational Site, Dunkirk
  - GSK Investigational Site, Fourmies
  - GSK Investigational Site, Grande-Synthe
  - GSK Investigational Site, Guilherand-Granges
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Le Raincy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Longjumeau
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Orsay
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pau
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Ploemeur
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Cyr-sur-Loire
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Grégoire
  - GSK Investigational Site, Saint-Martin-d'Hères
  - GSK Investigational Site, Saint-Nazaire
  - GSK Investigational Site, Saint-Quentin
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Troyes
  - GSK Investigational Site, Vannes
- Germany (146):
  - GSK Investigational Site, Backnang, Baden-Wurttemberg
  - GSK Investigational Site, Bad Schönborn, Baden-Wurttemberg
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Esslingen am Neckar, Baden-Wurttemberg
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Kleinblittersdorf, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Neckargemünd, Baden-Wurttemberg
  - GSK Investigational Site, Ostfildern, Baden-Wurttemberg
  - GSK Investigational Site, Rheinfelden, Baden-Wurttemberg
  - GSK Investigational Site, Waldkirch, Baden-Wurttemberg
  - GSK Investigational Site, Aichach, Bavaria
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Bad Griesbach, Bavaria
  - GSK Investigational Site, Bamberg, Bavaria
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Ebersberg, Bavaria
  - GSK Investigational Site, Forchheim, Bavaria
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Garmisch-Partenkirchen, Bavaria
  - GSK Investigational Site, Günzburg, Bavaria
  - GSK Investigational Site, Herzogenaurach, Bavaria
  - GSK Investigational Site, Höchberg, Bavaria
  - GSK Investigational Site, Kelheim, Bavaria
  - GSK Investigational Site, Koenigsbrunn, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Neumarkt in der Oberpfalz, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Planegg, Bavaria
  - GSK Investigational Site, Rosenheim, Bavaria
  - GSK Investigational Site, Roth, Bavaria
  - GSK Investigational Site, Starnberg, Bavaria
  - GSK Investigational Site, Weiden, Bavaria
  - GSK Investigational Site, Weißenburg in Bayern, Bavaria
  - GSK Investigational Site, Wertheim, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Hennigsdorf, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Schwedt, Brandenburg
  - GSK Investigational Site, Senftenberg, Brandenburg
  - GSK Investigational Site, Strausberg, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Wedel, Hamburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hochheim am Main, Hesse
  - GSK Investigational Site, Kelkheim, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Neustadt, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Seligenstadt, Hesse
  - GSK Investigational Site, Vellmar, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Braunschweig, Lower Saxony
  - GSK Investigational Site, Bremervörde, Lower Saxony
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Buxtehude, Lower Saxony
  - GSK Investigational Site, Ganderkesee, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Holzminden, Lower Saxony
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfsburg, Lower Saxony
  - GSK Investigational Site, Bad Doberan, Mecklenburg-Vorpommern
  - GSK Investigational Site, Ludwigslust, Mecklenburg-Vorpommern
  - GSK Investigational Site, Ribnitz-Damgarten, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Arnsberg, North Rhine-Westphalia
  - GSK Investigational Site, Bocholt, North Rhine-Westphalia
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Borken, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Dülmen, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Kamp-Lintfort, North Rhine-Westphalia
  - GSK Investigational Site, Kempen, North Rhine-Westphalia
  - GSK Investigational Site, Königswinter, North Rhine-Westphalia
  - GSK Investigational Site, Krefeld, North Rhine-Westphalia
  - GSK Investigational Site, Langenfeld, North Rhine-Westphalia
  - GSK Investigational Site, Marl, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Mülheim, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Paderborn, North Rhine-Westphalia
  - GSK Investigational Site, Pulheim, North Rhine-Westphalia
  - GSK Investigational Site, Wesseling, North Rhine-Westphalia
  - GSK Investigational Site, Wuppertal, North Rhine-Westphalia
  - GSK Investigational Site, Bad Bergzaben, Rhineland-Palatinate
  - GSK Investigational Site, Bad Ems, Rhineland-Palatinate
  - GSK Investigational Site, Dierdorf, Rhineland-Palatinate
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Nieder-Olm, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Bad Schlema, Saxony
  - GSK Investigational Site, Bautzen, Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Grimma, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Markkleeberg, Saxony
  - GSK Investigational Site, Neustadt, Saxony
  - GSK Investigational Site, Oelsnitz, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Plauen, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Schwarzenberg, Saxony
  - GSK Investigational Site, Wilkau-Haßlau, Saxony
  - GSK Investigational Site, Zwickau, Saxony
  - GSK Investigational Site, Dessau, Saxony-Anhalt
  - GSK Investigational Site, Eisleben Lutherstadt, Saxony-Anhalt
  - GSK Investigational Site, Gardelegen, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Leuna, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Naumburg, Saxony-Anhalt
  - GSK Investigational Site, Weißenfels, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Ahrensburg, Schleswig-Holstein
  - GSK Investigational Site, Bad Schwartau, Schleswig-Holstein
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Hemmoor, Schleswig-Holstein
  - GSK Investigational Site, Husum, Schleswig-Holstein
  - GSK Investigational Site, Itzehoe, Schleswig-Holstein
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lauenburg, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Plön, Schleswig-Holstein
  - GSK Investigational Site, Schleswig, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Gotha, Thuringia
  - GSK Investigational Site, Ilmenau, Thuringia
  - GSK Investigational Site, Meiningen, Thuringia
  - GSK Investigational Site, Waltershausen, Thuringia
- Greece (8):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Periohi Dragana, Alexandroupolis
  - GSK Investigational Site, Rhodes
  - GSK Investigational Site, Rio, Patras
  - GSK Investigational Site, Thessaloniki
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Miskolc
- Ireland (3):
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Tallaght
- Italy (15):
  - GSK Investigational Site, Lanciano (CH), Abruzzo
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Caserta, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Forlì, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Voghera (PV), Lombardy
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Ragusa (CT), Sicily
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Isola Della Scala (VR), Veneto
  - GSK Investigational Site, Napoli, Veneto
- Japan (6):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Ōita
- Latvia (2):
  - GSK Investigational Site, Daugavpils
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Šiauliai
  - GSK Investigational Site, Vilnius
- Mexico (6):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
  - GSK Investigational Site, Puebla City
- Netherlands (17):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Capelle aan den IJssel
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Roermond
  - GSK Investigational Site, Roosendaal
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Stadskanaal
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
- New Zealand (6):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Nelson
  - GSK Investigational Site, Tauranga
  - GSK Investigational Site, Whangarei
- Norway (5):
  - GSK Investigational Site, Arendal
  - GSK Investigational Site, Moelv
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Porsgrunn
  - GSK Investigational Site, Stavanger
- Poland (14):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Chęciny
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kościerzyna
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wejherowo
  - GSK Investigational Site, Wroclaw
- Portugal (4):
  - GSK Investigational Site, Almada
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Puerto Rico (2):
  - GSK Investigational Site, Ponce, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico
- GSK Investigational Site, Bucharest, Romania
- Russia (4):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Martin
- Slovenia (4):
  - GSK Investigational Site, Celje
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Maribor
  - GSK Investigational Site, Slovenj Gradec
- South Africa (8):
  - GSK Investigational Site, Rosebank, Gauteng
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Capital Park
  - GSK Investigational Site, George
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Parktown
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Westville, Durban
- Spain (31):
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Alcala de Henares (Madrid)
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Don Benito (Badajoz)
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Ibiza Town
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, La Laguna (Santa Cruz de Tenerife)
  - GSK Investigational Site, Leganés
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manacor
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Orihuela
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Sagunto
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Soria
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Via-Real (Castellón)
- Sweden (13):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gävle
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Karlshamn
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Skärholmen
  - GSK Investigational Site, Skövde
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Vålberg
- Switzerland (9):
  - GSK Investigational Site, Aarau
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Biel
  - GSK Investigational Site, Fribourg
  - GSK Investigational Site, Geneva
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Olten
  - GSK Investigational Site, Sarnen
  - GSK Investigational Site, Zollikon
- Tunisia (3):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Turkey (Türkiye) (4):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Capa/Istanbul
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Izmir
- Ukraine (4):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Zaporizhzhya
- United Kingdom (44):
  - GSK Investigational Site, Aberdeen, Aberdeenshire
  - GSK Investigational Site, Ayr, Ayrshire
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Stockport, Cheshire
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Bristol, Gloucestershire
  - GSK Investigational Site, Portsmouth, Hampshire
  - GSK Investigational Site, Southampton, Hampshire
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Lancs, Lancashire
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Oldham, Lancashire
  - GSK Investigational Site, Leicester, Leicestershire
  - GSK Investigational Site, Leytonstone, London
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Norwich, Norfolk
  - GSK Investigational Site, Newcastle upon Tyne, Northumberland
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Bath, Somerset
  - GSK Investigational Site, Tauton, Somerset
  - GSK Investigational Site, Stoke-on-Trent, Staffordshire
  - GSK Investigational Site, Redhill, Surrey
  - GSK Investigational Site, Chichester, Sussex West
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, Coventry, Warwickshire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Clydebank, Glasgow
  - GSK Investigational Site, Crewe
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, Falkirk
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Sheffield
  - GSK Investigational Site, Torquay
  - GSK Investigational Site, Wakefield
  - GSK Investigational Site, Waterloo, Liverpool
  - GSK Investigational Site, Wolverhampton
- GSK Investigational Site

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kader AK, Sun J, Reck BH, Newcombe PJ, Kim ST, Hsu FC, D'Agostino RB Jr, Tao S, Zhang Z, Turner AR, Platek GT, Spraggs CF, Whittaker JC, Lane BR, Isaacs WB, Meyers DA, Bleecker ER, Torti FM, Trent JM, McConnell JD, Zheng SL, Condreay LD, Rittmaster RS, Xu J. Potential impact of adding genetic markers to clinical parameters in predicting prostate biopsy outcomes in men following an initial negative biopsy: findings from the REDUCE trial. Eur Urol. 2012 Dec;62(6):953-61. doi: 10.1016/j.eururo.2012.05.006. Epub 2012 May 12. PMID 22652152
- [Background] Aubin SM, Reid J, Sarno MJ, Blase A, Aussie J, Rittenhouse H, Rittmaster R, Andriole GL, Groskopf J. PCA3 molecular urine test for predicting repeat prostate biopsy outcome in populations at risk: validation in the placebo arm of the dutasteride REDUCE trial. J Urol. 2010 Nov;184(5):1947-52. doi: 10.1016/j.juro.2010.06.098. Epub 2010 Sep 17. PMID 20850153
- [Background] Wu C, Moreira DM, Gerber L, Rittmaster RS, Andriole GL, Freedland SJ. Diabetes and prostate cancer risk in the REDUCE trial. Prostate Cancer Prostatic Dis. 2011 Dec;14(4):326-31. doi: 10.1038/pcan.2011.28. Epub 2011 Jun 28. PMID 21709690
- [Background] Roehrborn CG, Nickel JC, Andriole GL, Gagnier RP, Black L, Wilson TH, Rittmaster RS. Dutasteride improves outcomes of benign prostatic hyperplasia when evaluated for prostate cancer risk reduction: secondary analysis of the REduction by DUtasteride of prostate Cancer Events (REDUCE) trial. Urology. 2011 Sep;78(3):641-6. doi: 10.1016/j.urology.2011.03.063. Epub 2011 Jul 20. PMID 21764428
- [Background] Bostwick DG, Qian J, Drewnowska K, Varvel S, Bostwick KC, Marberger M, Rittmaster RS. Prostate needle biopsy quality in reduction by dutasteride of prostate cancer events study: worldwide comparison of improvement with investigator training and centralized laboratory processing. Urology. 2010 Jun;75(6):1406-10. doi: 10.1016/j.urology.2009.07.1348. Epub 2009 Nov 25. PMID 19942263
- [Background] Crawford ED, Andriole GL, Marberger M, Rittmaster RS. Reduction in the risk of prostate cancer: future directions after the Prostate Cancer Prevention Trial. Urology. 2010 Mar;75(3):502-9. doi: 10.1016/j.urology.2009.05.099. Epub 2009 Dec 29. PMID 20035983
- [Background] G Andriole, D Bostwick, O Brawley, L Gomella, M Marberger, F Montorsi, C Pettaway, T Tammela, C Teloken, D Tindall, M Somerville, I Fowler and R Rittmaster on behalf of the REDUCE Study Group. Risk reduction in men at increased risk: outcomes of the REduction by Dutasteride of prostate Cancer Events (REDUCE) trial. [N Engl J Med]. 2010;362(13):1192-202.
- [Background] Andriole GL, Bostwick D, Brawley OW, Gomella L, Marberger M, Montorsi F, Pettaway C, Tammela TL, Teloken C, Tindall D, Freedland SJ, Somerville MC, Wilson TH, Fowler I, Castro R, Rittmaster RS; REDUCE Study Group. The effect of dutasteride on the usefulness of prostate specific antigen for the diagnosis of high grade and clinically relevant prostate cancer in men with a previous negative biopsy: results from the REDUCE study. J Urol. 2011 Jan;185(1):126-31. doi: 10.1016/j.juro.2010.09.011. Epub 2010 Nov 12. PMID 21074214
- [Background] Andriole GL, Bostwick DG, Brawley OW, Gomella LG, Marberger M, Montorsi F, Pettaway CA, Tammela TL, Teloken C, Tindall DJ, Somerville MC, Wilson TH, Fowler IL, Rittmaster RS; REDUCE Study Group. Effect of dutasteride on the risk of prostate cancer. N Engl J Med. 2010 Apr 1;362(13):1192-202. doi: 10.1056/NEJMoa0908127. PMID 20357281
- [Background] Nickel JC, Roehrborn C, Montorsi F, Wilson TH, Rittmaster RS. Dutasteride reduces prostatitis symptoms compared with placebo in men enrolled in the REDUCE study. J Urol. 2011 Oct;186(4):1313-8. doi: 10.1016/j.juro.2011.05.071. Epub 2011 Aug 17. PMID 21849186
- [Background] Jean-Alfred Thomas, II, Leah Gerber, Lionel Banez, Daniel Moreira,Ramiro Castro, Gerald L. Andriole and Stephen J. Freedland. Prostate Cancer Risk in Men with Prostate and Breast Cancer Family History: Results from the REDUCE study. [J Intern Med [Epub Dec 28 2011]]. 2011;
- [Background] Marberger M, McConnell JD, Fowler I, Andriole GL, Bostwick DG, Somerville MC, Rittmaster RS. Biopsy misidentification identified by DNA profiling in a large multicenter trial. J Clin Oncol. 2011 May 1;29(13):1744-9. doi: 10.1200/JCO.2010.32.1646. Epub 2011 Mar 28. PMID 21444877
- [Background] Marberger M, Freedland SJ, Andriole GL, Emberton M, Pettaway C, Montorsi F, Teloken C, Rittmaster RS, Somerville MC, Castro R. Usefulness of prostate-specific antigen (PSA) rise as a marker of prostate cancer in men treated with dutasteride: lessons from the REDUCE study. BJU Int. 2012 Apr;109(8):1162-9. doi: 10.1111/j.1464-410X.2011.10373.x. Epub 2011 Jun 23. PMID 21699645
- [Background] Marberger M, Wilson TH, Rittmaster RS. Low serum testosterone levels are poor predictors of sexual dysfunction. BJU Int. 2011 Jul;108(2):256-62. doi: 10.1111/j.1464-410X.2010.09766.x. Epub 2010 Oct 18. PMID 20955266
- [Background] Kattan MW, Earnshaw SR, McDade CL, Black LK, Andriole GL. Cost effectiveness of chemoprevention for prostate cancer with dutasteride in a high-risk population based on results from the REDUCE clinical trial. Appl Health Econ Health Policy. 2011 Sep 1;9(5):305-15. doi: 10.2165/11592200-000000000-00000. PMID 21875161
- [Background] Muller RL, Gerber L, Moreira DM, Andriole G, Castro-Santamaria R, Freedland SJ. Serum testosterone and dihydrotestosterone and prostate cancer risk in the placebo arm of the Reduction by Dutasteride of Prostate Cancer Events trial. Eur Urol. 2012 Nov;62(5):757-64. doi: 10.1016/j.eururo.2012.05.025. Epub 2012 May 18. PMID 22658758
- [Background] Newcombe PJ, Reck BH, Sun J, Platek GT, Verzilli C, Kader AK, Kim ST, Hsu FC, Zhang Z, Zheng SL, Mooser VE, Condreay LD, Spraggs CF, Whittaker JC, Rittmaster RS, Xu J. A comparison of Bayesian and frequentist approaches to incorporating external information for the prediction of prostate cancer risk. Genet Epidemiol. 2012 Jan;36(1):71-83. doi: 10.1002/gepi.21600. PMID 22890972
- [Background] Aubin SM, Reid J, Sarno MJ, Blase A, Aussie J, Rittenhouse H, Rittmaster RS, Andriole GL, Groskopf J. Prostate cancer gene 3 score predicts prostate biopsy outcome in men receiving dutasteride for prevention of prostate cancer: results from the REDUCE trial. Urology. 2011 Aug;78(2):380-5. doi: 10.1016/j.urology.2011.03.033. PMID 21820580
- [Background] Stephen J. Freedland, Leah Gerber, Lionel Banez, Daniel Moreira, Gerald L. Andriole, and Roger S. Rittmaster on behalf of the REDUCE Study Group. Statin Use and the Risk of Prostate Cancer and High-grade Prostate Cancer: Results from the REDUCE study. [AUA 2011 Annual Meeting]. 2011;185(4 Suppl):e135.
- [Background] Thomas JA 2nd, Gerber L, Banez LL, Moreira DM, Rittmaster RS, Andriole GL, Freedland SJ. Prostate cancer risk in men with baseline history of coronary artery disease: results from the REDUCE Study. Cancer Epidemiol Biomarkers Prev. 2012 Apr;21(4):576-81. doi: 10.1158/1055-9965.EPI-11-1017. Epub 2012 Feb 7. PMID 22315364
- [Derived] Vidal AC, Oyekunle T, Feng T, Freedland AR, Moreira D, Castro-Santamaria R, Andriole GL, Freedland SJ, Allott EH. Asian Race and Risk of Prostate Cancer: Results from the REDUCE Study. Cancer Epidemiol Biomarkers Prev. 2020 Nov;29(11):2165-2170. doi: 10.1158/1055-9965.EPI-20-0646. Epub 2020 Aug 20. PMID 32856605
- [Derived] Bliwise DL, Howard LE, Moreira DM, Andriole GL, Hopp ML, Freedland SJ. Nocturia and associated mortality: observational data from the REDUCE trial. Prostate Cancer Prostatic Dis. 2019 Mar;22(1):77-83. doi: 10.1038/s41391-018-0090-5. Epub 2018 Sep 13. PMID 30214036
- [Derived] Moreira DM, Andriole GL, Nickel JC, Roehrborn CG, Castro-Santamaria R, Freedland SJ. Dutasteride is associated with reduced risk of transrectal prostate biopsy-associated urinary tract infection and related hospitalizations. World J Urol. 2017 Oct;35(10):1525-1530. doi: 10.1007/s00345-017-2036-2. Epub 2017 Apr 10. PMID 28396999
- [Derived] Nickel JC, Roehrborn CG, Castro-Santamaria R, Freedland SJ, Moreira DM. Chronic Prostate Inflammation is Associated with Severity and Progression of Benign Prostatic Hyperplasia, Lower Urinary Tract Symptoms and Risk of Acute Urinary Retention. J Urol. 2016 Nov;196(5):1493-1498. doi: 10.1016/j.juro.2016.06.090. Epub 2016 Jul 1. PMID 27378134
- [Derived] Moreira DM, Nickel JC, Andriole GL, Castro-Santamaria R, Freedland SJ. Chronic baseline prostate inflammation is associated with lower tumor volume in men with prostate cancer on repeat biopsy: Results from the REDUCE study. Prostate. 2015 Sep;75(13):1492-8. doi: 10.1002/pros.23041. Epub 2015 Jul 17. PMID 26184556
- [Derived] Moreira DM, Bostwick DG, Andriole GL, Peterson BL, Cohen HJ, Castro-Santamaria R, Freedland SJ. Baseline Prostate Atrophy is Associated with Reduced Risk of Prostate Cancer in Men Undergoing Repeat Prostate Biopsy. J Urol. 2015 Nov;194(5):1241-6. doi: 10.1016/j.juro.2015.05.103. Epub 2015 Jul 10. PMID 26165588
- [Derived] Toren P, Margel D, Kulkarni G, Finelli A, Zlotta A, Fleshner N. Effect of dutasteride on clinical progression of benign prostatic hyperplasia in asymptomatic men with enlarged prostate: a post hoc analysis of the REDUCE study. BMJ. 2013 Apr 15;346:f2109. doi: 10.1136/bmj.f2109. PMID 23587564
- [Derived] Muller RL, Gerber L, Moreira DM, Andriole G Jr, Hamilton RJ, Fleshner N, Parsons JK, Freedland SJ. Obesity is associated with increased prostate growth and attenuated prostate volume reduction by dutasteride. Eur Urol. 2013 Jun;63(6):1115-21. doi: 10.1016/j.eururo.2013.02.038. Epub 2013 Mar 7. PMID 23541458
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARI40006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo, repeat oral once daily dosing for 4 years. Placebo supplied as matching dutasteride capsules.
- Dutasteride 0.5 mg: Dutasteride 0.5 milligrams (mg), repeat oral once daily dosing for 4 years. Dutasteride supplied as gelatin capsule.
Period: Overall Study
Arm/Group | Placebo | Dutasteride 0.5 mg
Started | 4126 | 4105
Completed | 2915 | 2912
Not Completed | 1211 | 1193
Not completed — Adverse Event | 282 | 364
Not completed — Withdrawal by Subject | 377 | 361
Not completed — Lost to Follow-up | 123 | 113
Not completed — Protocol Violation | 104 | 95
Not completed — Diagnosed with Prostate Cancer | 202 | 166
Not completed — Listed as "Other" on Case Report Form | 98 | 60
Not completed — Missing | 25 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dutasteride 0.5 mg | Total
Number analyzed (Participants) | 4126 | 4105 | 8231
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (6.08) | 62.8 (6.04) | 62.8 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4126 | 4105 | 8231
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3747 | 3744 | 7491
  Black | 99 | 91 | 190
  Asian | 67 | 67 | 134
  American Hispanic | 173 | 160 | 333
  Other | 39 | 43 | 82
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biopsy-detectable Prostate Cancer at Years 2 and 4 (Crude Rate Approach)
Description: Study biopsies consisted of 10 biopsy samples (cores) in a pre-defined pattern. Biopsies were read at the central pathology laboratory (CPL, which processed the majority, 94%, of biopsies). Biopsy cases that were positive for prostate cancer or precancerous lesions (high-grade prostatic intraepithelial neoplasia[HGPIN] or typical small acinar proliferation [ASAP]) and prostate surgeries were reviewed by the lead pathologist.
Time Frame: Years 1-2, Years 3-4, and Overall (Years 1-4)
Population: Efficacy Population: all randomized participants with a negative entry biopsy, as determined by the CPL, who received at least 1 dose of study drug. The crude rate approach included all participants at risk at the beginning of each time period .
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants
  Years 1- 2, n=4073, 4049 | 578 | 435
  Years 3- 4, n=2815, 2844 | 280 | 224
  Overall, n=4073, 4049 | 858 | 659
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.0001, Mantel-Cox — The p value is given is for the overall assessment; Relative Risk Reduction = 23.3, 95% CI [15.6 to 30.3] — Estimation data given are for the overall assessment

2. Primary Outcome: Number of Participants With Biopsy-detectable Prostate Cancer at Years 2 and 4 (Modified Crude Rate Approach)
Description: Study biopsies (biop.) consisted of 10 biop. samples (cores) in a pre-defined pattern and were read at the central pathology laboratory. Biop. cases that were positive for prostate cancer or precancerous lesions (HGPIN or ASAP) and prostate surgeries were reviewed by the lead pathologist. Participants included in the risk sets at Years 1-2 and Years 3-4 included those with a positive biop. at Years 1-2 or a biop. after Months 18-24, and those with a positive biop. at Years 3-4 or a biop. after Month 42, respectively. Overall included participants with a positive biop. or biop. after Month 42.
Time Frame: Years 1-2, Years 3-4, and Overall (Years 1-4)
Population: Efficacy Population, modified crude rate: participants who either were diagnosed with prostate cancer during the study or had an end of time period biopsy. N for each time period is the number who either had at least 1 biopsy in the final 6 months of the time period or had a positive biopsy anytime during the time period.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3319 | 3209
participants
  Years 1-2, n=3319, 3209 | 578 | 435
  Years 3-4, n=2325, 2434 | 280 | 224
  Overall, n=2903, 2869 | 858 | 659
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.0001, Mantel-Cox — The p value is given is for the overall assessment; Relative Risk Reduction = 23.1, 95% CI [15.5 to 30.0] — Estimation data are given are for the overall assessment

3. Primary Outcome: Number of Participants With Biopsy-detectable Prostate Cancer at Years 2 and 4 (Restricted Crude Rate Approach)
Description: Study biopsies consisted of 10 biopsy samples (cores) in a pre-defined pattern. Biopsies were read at the central pathology laboratory (which processed the majority, 94%, of biopsies). Biopsy cases that were positive for prostate cancer or precancerous lesions (HGPIN or ASAP) and prostate surgeries were reviewed by the lead pathologist. Participants included in the risk set at Years 1-2, Years 3-4, and Overall (Years 1-4) were those who had a biopsy during the specified time period.
Time Frame: Years 1-2, Years 3-4, and Overall (Years 1-4)
Population: Efficacy Population, restricted crude rate: the number of prostate cancer events is based on the the number of participants who had at least one biopsy during the time period. Ns at Years 1-2 and Years 3-4 are the number who had a biopsy in those time periods; the overall n is the number of participants who had 1 or more biopsy during Years 1-4.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3424 | 3305
participants
  Years 1-2, n=3364, 3244 | 578 | 435
  Years 3- 4, n=2359, 2451 | 280 | 224
  Overall, n=3424, 3305 | 858 | 659
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.0001, Mantel-Cox — The p value is given for the overall assessment; Relative Risk Reduction = 22.8, 95% CI [15.2 to 29.8] — Estimation data are given for the overall assessment

4. Secondary Outcome: Number of Participants With the Indicated Gleason Score at Diagnosis
Description: Gleason score was determined by examining prostate biopsies and surgical samples. The Gleason scoring system sums the two most common Gleason grade patterns in order to predict the likelihood of a participant doing well or badly with their cancer. Gleason grades range from 1 (normal) to 5 (advanced cancer). The lowest Gleason score is 2 (1+1), and the highest Gleason score is 10 (5+5). A Gleason score of 2-6 is a low-grade cancer; a Gleason score of 7-10 is high-grade cancer. The most severe high-grade cancers are the subset of Gleason scores 8-10.
Time Frame: Baseline to Year 4
Population: Biopsied Population: all randomized participants with a negative entry biopsy who received at least 1 dose of study treatment and who had at least 1 biopsy reviewed by the central pathology lab. Only needle biopsies are included (surgeries are excluded). The number analyzed is smaller than the total number in the population due to missing values.
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3407 | 3299
participants
  Between 2 and 6 | 617 | 437
  Between 7 and 10 | 233 | 220
  Between 8 and 10 | 19 | 29

5. Secondary Outcome: Number of Participants With HGPIN, ASAP, and Prostate Cancer at Biopsy
Description: The occurrence and quantity of high-grade prostatic intraepithelial neoplasia (HGPIN) and atypical small acinar proliferation (ASAP) at biopsy were measured. HGPIN and ASAP are considered precancerous conditions. A participant diagnosed with prostate cancer only (i.e., no HGPIN or ASAP) was counted in both the first category ("HGPIN or prostate cancer diagnosis") and again in the last category ("HGPIN, ASAP, or prostate cancer diagnosis").
Time Frame: Baseline to Year 4
Population: Biopsied Population: the number analyzed is the total number in the population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3424 | 3305
participants
  HGPIN or prostate cancer diagnosis | 1126 | 810
  HGPIN and no prostate cancer | 268 | 151
  HGPIN and no ASAP and no prostate cancer | 206 | 121
  HGPIN or ASAP | 675 | 409
  HGPIN or ASAP and no prostate cancer | 373 | 248
  HGPIN, ASAP, or prostate cancer diagnosis | 1231 | 907

6. Secondary Outcome: Volume of HGPIN at Biopsy
Description: The amount of prostate biopsy tissue with HGPIN was measured.
Time Frame: Baseline to Year 4
Population: Biopsied Population. Only needle biopsies are included (surgeries are excluded). The number analyzed is smaller than the total number in the population due to missing values.
Measure: Mean (Standard Deviation); unit: cc*10^-3 (microliter)
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3403 | 3297
cc*10^-3 (microliter) | 0.1105 (0.52753) | 0.0446 (0.2771)

7. Secondary Outcome: Percentage of Core Involved at Diagnosis
Description: The average amount of cancer seen by the pathologist in the prostate tissue samples taken during the biopsy was measured. A core is a prostate biopsy sample.
Time Frame: Baseline to Year 4
Population: Prostate Cancer Population: all participants in the Efficacy Population who received a post-baseline diagnosis of prostate cancer by the central pathology laboratory. Only needle biopsies are included (surgeries are excluded). The number analyzed is smaller than the total number in the population due to missing values.
Measure: Mean (Standard Deviation); unit: percentage of core
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 849 | 657
percentage of core | 13.4 (14.84) | 12.2 (13.00)

8. Secondary Outcome: Number of Cancer-positive Cores
Description: The average number of prostate biopsy samples (cores) determined to be cancerous by the pathologist was measured. Normally, 10 cores were taken per biopsy for each participant.
Time Frame: Baseline to Year 4
Population: Prostate Cancer Population. Only needle biopsies are included (surgeries are excluded). The number analyzed is smaller than the total number in the population due to missing values.
Measure: Mean (Standard Deviation); unit: number of cores
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 850 | 656
number of cores | 1.9 (1.31) | 1.8 (1.33)

9. Secondary Outcome: Treatment Alteration Score
Description: The treatment alteration score is a measure of the cellular changes due to treatment (effect of male hormone withdrawal) on the nucleus and cytoplasm of the prostate cancer cell. The treatment alteration score is the sum of two scores (the nuclear alteration score and the cytoplasmic architectural score), each ranging from 0 to 3, with 0 indicating no change and 3 indicating severe changes.
Time Frame: Baseline to Year 4
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3357 | 3258
points on a scale
  Nuclear, n=3357, 3256 | 0.008 (0.1116) | 0.019 (0.1734)
  Architectural, n=3357, 3258 | 0.009 (0.1289) | 0.023 (0.2112)
  Total, n=3357, 3256 | 0.017 (0.2336) | 0.041 (0.3737)

10. Secondary Outcome: Number of Participants Undergoing Intervention (Surgical and Non-surgical) for Prostate Cancer Treatment
Description: The number of participants who received treatment for prostate cancer was measured. Prostate cancer interventions included surgical interventions (e.g., prostatectomy, adenomectomy, transurethral resection) and non-surgical interventions (e.g., chemotherapy, hormone therapy, radiation therapy).
Time Frame: Baseline to Year 4
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants
  Any intervention | 438 | 300
  Any surgical intervention | 304 | 221
  Any non-surgical intervention | 172 | 95

11. Secondary Outcome: Adjusted Mean Change From Baseline in the International Prostate Symptom Score (IPSS) at Month 48
Description: The IPSS is a 7-item questionnaire that measures urinary symptoms. It measures the level of urinary symptoms (including incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) reported as the total IPSS score. Each of the 7 questions has a 6-point response scale (0=none/not at all to 5=almost always) with a total score that can range from 0-35: mild (0-7), moderate (8-19), or severe (20-35). Estimates are based on adjusted means from the general linear model: change from baseline = baseline value and cluster and treatment.
Time Frame: Baseline to Year 4 (Month 48)
Population: Efficacy Population, last observation carried forward (LOCF). In the LOCF approach, missing values at post-baseline assessments are replaced with the participant's previous non-missing post-baseline assessment. The number analyzed is smaller than the total number in the population due to missing values.
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3847 | 3815
points on a scale | 1.35 (0.087) | -0.46 (0.087)

12. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in Prostate Volume at Months 24 and 48
Description: Prostate volume was measured by transrectal ultrasound (TRUS) when biopsies were performed at Year 2 and Year 4. The investigator calculated the prostate volume using three prostate measurements (anteroposterior, cephalocaudal, and transverse diameters). Estimates are based on the adjusted means from the general linear model: log(Post-Baseline/Baseline value) = treatment and cluster and log (baseline value).
Time Frame: Baseline, Month 24, and Month 48
Population: Efficacy Population (LOCF). The number analyzed is smaller than the total number in the population due to missing values.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3289 | 3194
percent change
  Month 24, n=3192, 3116 | 13.0 (0.65) | -17.4 (0.48)
  Month 48, n=3289, 3194 | 19.7 (0.77) | -17.5 (0.54)

13. Secondary Outcome: Adjusted Mean Change From Baseline in Maximum Urinary Flow (Qmax) at Months 12, 24, 36, and 48
Description: Maximum urinary flow was measured at selected sites using a Dantec Uroflow meter with a Thompson filter. Change from baseline was calculated as Month 12, 24, 36, and 48 values minus the baseline value. Estimates are based on the adjusted means from the general linear model: change from baseline = baseline Qmax and treatment. This measurement was performed at selected centers.
Time Frame: Baseline and Months 12, 24, 36, and 48
Population: as for outcome 12
Measure: Mean (Standard Error); unit: milliliters/second
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 1390 | 1359
milliliters/second
  Month 12, n=1178, 1168 | -0.55 (0.253) | 0.27 (0.255)
  Month 24, n=1337, 1295 | -0.63 (0.410) | 0.60 (0.416)
  Month 36, n=1375, 1334 | -0.74 (0.238) | 0.13 (0.241)
  Month 48, n=1390, 1359 | -0.90 (0.303) | 0.41 (0.307)

14. Secondary Outcome: Number of Participants Starting Alpha Blockers to Control Benign Prostatic Hyperplasia (BPH) Symptoms
Description: Medication taken during the study, including alpha blockers, was recorded at each 6-month study visit and during phone calls that occurred 3 months after each visit.
Time Frame: Years 1-2, Overall (Years 1-4)
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants
  Years 1-2 | 425 | 317
  Overall | 770 | 515

15. Secondary Outcome: Number of Participants With at Least One Event of Acute Urinary Retention (AUR)
Description: A participant was considered to have AUR when he reported being unable to urinate and required catherization. Participants were asked to report any events of AUR during the study.
Time Frame: Years 1-2 and Overall (Years 1-4)
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants
  Years 1-2 | 150 | 39
  Overall | 272 | 63

16. Secondary Outcome: Number of Participants With at Least One Urinary Tract Infection (UTI)
Description: A participant was considered to have a UTI if the investigator noted that the participant had UTI symptoms and had been prescribed antibiotics. Participants were asked to report any events of UTI during the study.
Time Frame: Years 1-2, Years 3-4, and Overall (Years 1-4)
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants
  Years 1-2, n=4073, 4049 | 196 | 131
  Years 3-4, n=3363, 3318 | 164 | 83
  Overall, n=4073, 4049 | 360 | 214

17. Secondary Outcome: Number of Participants With Post-biopsy Macroscopic Hematuria
Description: Participants reported events of macroscopic hematuria (visible blood in the urine) throughout the study.
Time Frame: Baseline to Year 4
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants | 168 | 127

18. Secondary Outcome: Number of Participants With Post-biopsy Macroscopic Hematospermia
Description: Participants reported events of macroscopic hematospermia (visible blood in semen) throughout the study.
Time Frame: Baseline through Year 4
Population: Efficacy Population
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
participants | 78 | 53

19. Secondary Outcome: Overall Survival
Description: Overall survival is assessed as the number of deaths reported throughout the study.
Time Frame: From time informed consent is signed to 4-month Safety Follow-Up period
Population: Efficacy Population
Measure: Number; unit: number of deaths
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 4073 | 4049
number of deaths
  Years 1-2 | 29 | 32
  Overall | 77 | 70

20. Secondary Outcome: Adjusted Mean Change From Baseline in the Benign Prostatic Hypertrophy (BPH) Impact Index (BII) at Month 48
Description: The BII is a 4-item questionnaire that rates the level of BPH-related physical discomfort, worry, and interference with normal activities the participant has experienced. The total BII score ranges from 1 (no impact on symptoms) to 13 (major impact on symptoms). Participants completed the questionnaire at Baseline and at each 6-month visit. Participants whose language did not have a validated translation of the questionnaire did not participate. Estimates are based on the adjusted means from the general linear model:change from baseline = baseline value and cluster and treatment.
Time Frame: Baseline and Month 48
Population: Efficacy Population (LOCF). The numbers presented are less than the overall population, as data were not available for all participants.
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3733 | 3727
points on a scale | 0.44 (0.037) | -0.21 (0.037)

21. Secondary Outcome: Adjusted Mean Change From Baseline in The Medical Outcomes Study Sleep Problems Index 6-item Standard Version (MOS Sleep-6S) at Month 48
Description: The MOS Sleep-6S is a 6-item questionnaire measuring quality of sleep. Scores range from 1 (all of the time) to 6 (none of the time) and are converted to a 1-100 scale and then averaged; a higher score indicates greater negative impact, which indicates more sleep disturbance. Participants completed the questionnaire at Baseline and at each 6-month visit. Participants whose language did not have a validated translation of the questionnaire did not participate. Estimates are based on the adjusted means from the general linear model: change from baseline=baseline value and cluster and treatment.
Time Frame: Baseline and Month 48
Population: as for outcome 20
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3726 | 3709
points on a scale | -0.03 (0.211) | 0.02 (0.212)

22. Secondary Outcome: Adjusted Mean Change From Baseline in the National Institutes of Health Chronic Prostatitis Symptom Index (NIH CPSI) at Month 48
Description: The NIH CSPI is a 9-item questionnaire that measures chronic prostatitis symptoms. The total score ranges from 0 to 43. A higher score indicates greater negative impact of prostatitis. Participants completed the questionnaire at Baseline and at each 6-month visit. Participants whose language did not have a validated translation of the questionnaire did not participate. Estimates are based on the adjusted means from the general linear model: change from Baseline = Baseline Value and Cluster and Treatment.
Time Frame: Baseline and Month 48
Population: as for outcome 20
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 2576 | 2590
points on a scale | 0.94 (0.123) | -0.37 (0.123)

23. Secondary Outcome: Adjusted Mean Change From Baseline in Quality of Life Question 8 (QOL Q8) at Month 48
Description: The QOL Q8 is the last question of the IPSS Questionnaire. It is a question about the participant's quality of life as it relates to prostate symptoms. Responses range from 0 (most positive) to 6 (most negative). A higher score indicates worse quality of life. Participants completed the questionnaire at Screening, Baseline, and at each 6-month visit. Estimates are based on the adjusted means from the general linear model: change from baseline = baseline value and cluster and treatment.
Time Frame: Baseline and Month 48
Population: as for outcome 12
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3853 | 3821
points on a scale | -0.06 (0.018) | -0.33 (0.018)

24. Secondary Outcome: Adjusted Mean Change From Baseline in the Problem Assessment Scale of the Sexual Function Index (PASSFI) at Month 48
Description: The PASSFI is a 3-item questionnaire that measures sexual function. Responses range from 0 (big problem) to 4 (no problem), with a total score of 12. A higher score indicates fewer problems with sexual functioning. Participants completed the questionnaire at Baseline and then yearly . Participants whose language did not have a validated translation of the questionnaire did not participate. Estimates are based on the adjusted means from the general linear model: change from baseline = baseline value and cluster and treatment.
Time Frame: Baseline and Month 48
Population: as for outcome 12
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3413 | 3329
points on a scale | -0.82 (0.064) | -1.5 (0.065)

25. Secondary Outcome: Number of Participants With the Indicated Serum Dihydrotestosterone (DHT) Concentration at Month 48
Description: Number of participants whose DHT, the active form of the male sex hormone testosterone, was less than 0.555 nanomoles/liter and below the level of detection at Month 48 was measured. It was measured by taking blood samples at screening and yearly thereafter.
Time Frame: Month 48
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3865 | 3822
participants
  <0.555 nanomoles/Liter | 493 | 3414
  <level of detection | 42 | 2210

26. Secondary Outcome: Mean Change From Baseline in Testosterone at Month 48
Description: Testosterone, a male sex hormone, was measured by taking blood samples at screening and yearly thereafter.
Time Frame: Baseline and Month 48
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride 0.5 mg
Number analyzed (Participants) | 3841 | 3796
percent change | -0.1 (36.95) | 20.0 (44.05)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride 0.5 mg; Test type: Superiority or Other; p < 0.001, general linear model, t-test; Difference in adjusted means = 18.8, 95% CI [17.3 to 20.4] — The adjusted mean difference was calculated as the difference between the adjusted means (-6.1 and 12.7) for the placebo and Dutasteride arms, respectively

ADVERSE EVENTS:
Arm/Group | Placebo | Dutasteride 0.5 mg
Serious Adverse Events (participants affected / at risk) | 837/4126 | 748/4105
Other Adverse Events (participants affected / at risk) | 1151/4126 | 1296/4105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4126) | Dutasteride 0.5 mg (N=4105)
Abdominal abscess (Infections and infestations) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 4 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 9 | 9
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 35 | 14
Angina unstable (Cardiac disorders) | 7 | 9
Aortic valve disease (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 2 | 1
Appendicitis (Infections and infestations) | 12 | 2
Arrhythmia (Cardiac disorders) | 16 | 6
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 3
Arthritis bacterial (Infections and infestations) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 21 | 18
Atrial flutter (Cardiac disorders) | 7 | 2
Atrial tachycardia (Cardiac disorders) | 2 | 0
Atrioventricular block (Cardiac disorders) | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 2 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bacteraemia (Infections and infestations) | 3 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Brain abscess (Infections and infestations) | 1 | 1
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 1
Candida sepsis (Infections and infestations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 6 | 1
Cardiac disorder (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 4 | 12
Cardiac failure acute (Cardiac disorders) | 1 | 3
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 7
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 4
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 3 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 5
Cholangitis suppurative (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic myelomonocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 11
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 2 | 6
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Coronary artery disease (Cardiac disorders) | 23 | 36
Coronary artery occlusion (Cardiac disorders) | 5 | 4
Coronary artery stenosis (Cardiac disorders) | 10 | 8
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Cystitis (Infections and infestations) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 3 | 2
Diverticulum (Gastrointestinal disorders) | 2 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dysplastic naevus syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Empyema (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Fibromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 4 | 9
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 2 | 1
Gastrointestinal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Gastrointestinal dysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 2 | 2
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Hepatitis E (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 3
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Infected bites (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 2
Infective tenosynoyitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 28 | 31
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Labyrinthitis (Infections and infestations) | 3 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 12
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningitis borrelia (Infections and infestations) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Mitral valve prolapse (Cardiac disorders) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Myocardial infarction (Cardiac disorders) | 43 | 38
Myocardial ischaemia (Cardiac disorders) | 5 | 7
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nosocomial infection (Infections and infestations) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Orchitis (Infections and infestations) | 4 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 4 | 3
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditits (Cardiac disorders) | 3 | 2
Peritonitis (Gastrointestinal disorders) | 1 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngoesophageal diverticulm (Gastrointestinal disorders) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 25 | 24
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Polyp colorectal (Gastrointestinal disorders) | 1 | 0
Post procedural infection (Infections and infestations) | 2 | 1
Post procedural sepsis (Infections and infestations) | 7 | 1
Postinfarction angina (Cardiac disorders) | 0 | 1
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 4 | 1
Proctocolitis (Gastrointestinal disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Prostate infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 1
Pulmonary valve stenosis (Cardiac disorders) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 6 | 4
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 17 | 3
Septic shock (Infections and infestations) | 2 | 1
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Sinoatrial block (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 2
Small intestinal perforation (Gastrointestinal disorders) | 0 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Streptococcal infection (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 3 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 4 | 1
Testicular abscess (Infections and infestations) | 2 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 2
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary tract infection (Infections and infestations) | 6 | 4
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 6 | 4
Ventricle rupture (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 2
Vestibular neuronitis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 2 | 0
Viral labyrinthitis (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Wound infection (Infections and infestations) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 19 | 22
Transient ischaemic attack (Nervous system disorders) | 13 | 8
Syncope (Nervous system disorders) | 6 | 9
Cerebral infarction (Nervous system disorders) | 2 | 5
Dizziness (Nervous system disorders) | 6 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 4
Epilepsy (Nervous system disorders) | 3 | 3
Cerebrovascular disorder (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 3 | 0
Presyncope (Nervous system disorders) | 1 | 2
Cartoid artery occlusion (Nervous system disorders) | 1 | 2
Lacunar infarction (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 1 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 1
Cerebral thrombosis (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1
Myasthenia gravis (Nervous system disorders) | 2 | 0
Myelopathy (Nervous system disorders) | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypertonia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Motor neurone disease (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Paresis (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1
Syringomyelia (Nervous system disorders) | 1 | 0
Temporal lobe epilepsy (Nervous system disorders) | 1 | 0
Arachnoid cyst (Nervous system disorders) | 1 | 0
Cartoid sinus syndrome (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Global amnesia (Nervous system disorders) | 1 | 0
Cluster headache (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 1 | 0
Cartoid artery disease (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Hemicephalalgia (Nervous system disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 8 | 7
Rib fracture (Injury, poisoning and procedural complications) | 2 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 6 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 4 | 4
Femur fracture (Injury, poisoning and procedural complications) | 4 | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 3 | 4
Fibula fracture (Injury, poisoning and procedural complications) | 5 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 4
Head injury (Injury, poisoning and procedural complications) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 3
Wound (Injury, poisoning and procedural complications) | 0 | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 3
Cartilige injury (Injury, poisoning and procedural complications) | 1 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2
Injury (Injury, poisoning and procedural complications) | 2 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 2
Scapula fracture (Injury, poisoning and procedural complications) | 2 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 2 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 1
Blast injury (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Adrenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Crush injury (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic coma (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 26 | 39
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6
Arthralgia (Metabolism and nutrition disorders) | 2 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 3 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 8
Deep vein thrombosis (Vascular disorders) | 8 | 6
Aortic aneurysm (Vascular disorders) | 5 | 5
Hypertensive crisis (Vascular disorders) | 3 | 4
Arteriosclerosis (Vascular disorders) | 1 | 3
Hypotension (Vascular disorders) | 3 | 1
Thrombophlebitis (Vascular disorders) | 1 | 3
Aortic stenosis (Vascular disorders) | 2 | 1
Haematoma (Vascular disorders) | 1 | 2
Intermittent claudication (Vascular disorders) | 1 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 3
Thrombosis (Vascular disorders) | 0 | 3
Varicose vein (Vascular disorders) | 3 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 1
Venous thrombosis (Vascular disorders) | 2 | 0
Aneurysm ruptured (Vascular disorders) | 2 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 1
Aortic rupture (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0
Aneurysm (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Iliac artery thrombosis (Vascular disorders) | 0 | 1
Labile blood pressure (Vascular disorders) | 1 | 0
Necrosis ischaemic (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Wound haemorrhage (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Venous occlusion (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
Aortic elongation (Vascular disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 17 | 3
Calculus ureteric (Renal and urinary disorders) | 5 | 11
Nephrolithiasis (Renal and urinary disorders) | 7 | 8
Haematuria (Renal and urinary disorders) | 9 | 3
Renal failure (Renal and urinary disorders) | 5 | 3
Renal colic (Renal and urinary disorders) | 3 | 4
Calculus bladder (Renal and urinary disorders) | 3 | 3
Renal failure acute (Renal and urinary disorders) | 3 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 3 | 1
Urethral stenosis (Renal and urinary disorders) | 3 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Extravasation of urine (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Urinoma (Renal and urinary disorders) | 0 | 1
Hyperuricosuria (Renal and urinary disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adenoidal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 10 | 16
Cholecystitis (Hepatobiliary disorders) | 6 | 6
Cholecystitis acute (Hepatobiliary disorders) | 7 | 5
Cholangitis (Hepatobiliary disorders) | 2 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 18 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 10 | 5
Epididymitis (Reproductive system and breast disorders) | 4 | 6
Prostatism (Reproductive system and breast disorders) | 2 | 0
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Peyronie's Disease (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Retrograde ejaculation (Reproductive system and breast disorders) | 0 | 1
Testicular cyst (Reproductive system and breast disorders) | 1 | 0
Genital discomfort (Reproductive system and breast disorders) | 0 | 1
Chest pain (General disorders) | 6 | 3
Non-cardiac chest pain (General disorders) | 4 | 4
Pyrexia (General disorders) | 3 | 4
Death (General disorders) | 2 | 1
Odema peripheral (General disorders) | 2 | 1
Chest discomfort (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Hernia obstructive (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 2
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Retinal detachment (Eye disorders) | 4 | 6
Glaucoma (Eye disorders) | 3 | 0
Cataract (Eye disorders) | 0 | 2
Retinal haemorrhage (Eye disorders) | 1 | 1
Retinal vein thrombosis (Eye disorders) | 2 | 0
Blindness (Eye disorders) | 1 | 0
Corneal opacity (Eye disorders) | 1 | 0
Maculopathy (Eye disorders) | 0 | 1
Myopia (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Retinal ischaemia (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0
Retinoschisis (Eye disorders) | 1 | 0
Depression (Psychiatric disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1
Mental change status (Psychiatric disorders) | 2 | 0
Mental disorder (Psychiatric disorders) | 0 | 2
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholic psychosis (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Impaired self-care (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Insulin-requiring Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 4 | 4
Phimosis (Congenital, familial and genetic disorders) | 2 | 2
Hip dysplasia (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 6
Labyrinthine fistula (Ear and labyrinth disorders) | 0 | 1
Vestibular ataxia (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Neurosensory hypoacusis (Ear and labyrinth disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Cardiac enzymes increased (Investigations) | 0 | 1
Full blood count abnormal (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Goitre (Endocrine disorders) | 3 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 1
Cushing's Syndrome (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Polyarteritis nodosa (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 0
Allergy to plants (Immune system disorders) | 0 | 1
Joint prosthesis user (Social circumstances) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4126) | Dutasteride 0.5 mg (N=4105)
Nasopharyngitis (Infections and infestations) | 288 | 313
Influenza (Infections and infestations) | 212 | 204
Erectile dysfunction (Reproductive system and breast disorders) | 363 | 494
Hypertension (Cardiac disorders) | 321 | 349
Back pain (Musculoskeletal and connective tissue disorders) | 245 | 261

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.